CLINICAL TRIAL: NCT02548598
Title: Analysis of Inflammation and Microbiome in Patients With Sinusitis and Asthma
Acronym: AIMS
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 14-14945
Record Dates: First submitted 2015-08-18; First posted 2015-09-14 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Asthma; Chronic Rhinosinusitis
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Mucus collected from the airway, induced sputum, brushings from the airway epithelium, mucus collected from the nasal passages, and blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- AIMS-Full Characterization: Participants in this group undergo characterization at the UCSF Airway Clinical Research Center 6 weeks following their scheduled sinus surgery.
  Interventions: Procedure: Endoscopic sinus surgery
- AIMS-OR: Participants in this group complete limited questionnaires and provide biological samples that are collected during their scheduled sinus surgery. No further characterization in done in this group.
  Interventions: Procedure: Endoscopic sinus surgery
- AIMS-M: Participants returning to UCSF Sinus Center clinic following sinus surgery who have nasal secretions that are removed by a study clinician will provide samples at these clinic visits.
  Interventions: Procedure: Endoscopic sinus surgery

INTERVENTIONS:
Procedure: Endoscopic sinus surgery — This is an observational trial of patients with and without asthma who have concomitant chronic rhinosinusitis requiring endoscopic sinus surgery.

SUMMARY:
This is a cross-sectional, non-interventional study, consisting of three study arms, (1) Full Characterization (AIMS-Full), (2) Surgery Arm (AIMS-OR), and (3) Mucus Collection (AIMS-M). Participants will be recruited and enrolled in either AIMS-Full or AIMS-OR (based on participant availability). Participants who complete the initial characterization study (either AIMS-Full or AIMS-OR), may also go on to participate in the AIMS-M arm, which focuses mainly on sample collection. Participants who choose not to participate in either characterization arm are able to enroll directly into AIMS-M for sample collection only.

DETAILED DESCRIPTION:
This is a cross-sectional and non-interventional study to investigate mechanisms of disease in patients with asthma who have concomitant chronic sinusitis and/or nasal polyps (upper airway disease). Approximately 160 participants will be enrolled. Patients who are scheduled to undergo inpatient or outpatient endoscopic sinus surgery at the University of California San Francisco for clinical management of their upper airway disease will be invited to participate. Leftover tissues or mucus from the surgery will be collected and processed for research purposes.

This study consists of three study arms, (1) Full Characterization (AIMS-Full), (2) Surgery (AIMS-OR), and (3) Mucus Collection (AIMS-M). Participants will be recruited and enrolled in either AIMS-Full or AIMS-OR (based on participant availability). Participants who complete the initial characterization study (either AIMS-Full or AIMS-OR), may also go on to participate in the AIMS-M arm, which focuses mainly on sample collection. Participants who choose not to participate in either characterization arm are able to enroll directly into AIMS-M for sample collection only.

Suitable patients, undergoing endoscopic sinus surgery, will be identified and recruited by the study team. Patients will first be asked to participate in the AIMS-Full characterization.

If patients are unable or unwilling to participate in AIMS-Full, they will have the option to take part in the AIMS-OR or AIMS-M arms.

AIMS-OR will consist of the endoscopic sinus surgery with an optional pre-procedure visit during which consent and blood specimens will be obtained and questionnaires will be administered. If the optional pre-procedure visit is not done, consent will be obtained at the surgery visit, and blood will not be collected.

AIMS-M will consist of up to 5 visits. Patients seen in the UCSF Sinus Center clinic may have clearance of sinus mucus as part of routine clinical care; AIMS-M visits will collect these mucus samples that would otherwise be discarded. Sinus mucus obtained at the clinic visit may be used for research purposes if patients have given consent to participate in the AIMS-M arm of the study.

Participants in all three study arms will complete study-specific questionnaires on asthma and allergy history and impairment and provide samples of nasal secretions that are collected as part of routine clinical care and would otherwise be discarded. Those participating in either characterization arm (AIMS-Full or AIMS-OR) will also provide nasal tissues (part of routine surgical procedure); airway epithelial brushings and blood collection (for study purposes only). Those participating in AIMS-Full will also participate in the following study procedures: medical history and physical exam (including vital signs and body anthropometrics), spirometry, methacholine challenge or airway reversibility testing, exhaled nitric oxide, questionnaires (asthma, sinusitis, metabolic health), urine collection, and sputum induction. A participant's time commitment to the study will vary depending on which arm the participant is enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age at Visit 0.
2. Diagnosis of bilateral chronic sinusitis with a minimum Lund-MacKay CT score of 6 and/or diagnosis of nasal polyps
3. Half of the patients need to have a history of asthma

Exclusion Criteria:

1. History of lung disease other than asthma (e.g., cystic fibrosis, chronic obstructive pulmonary disease, interstitial lung disease, etc.)
2. History of hiatal hernia repair
3. History of cigarette and/or marijuana smoking (>10 total pack years, smokes >5 cigarettes per month, smoking within 2 weeks of study participation, marijuana use within 1 month of study participation)
4. If a participant has had an upper respiratory tract infection and/or an exacerbation of his/her asthma within 4-6 weeks of the characterization visit, this visit will be rescheduled to 4 weeks after recovery.
5. Current pregnancy or breastfeeding
6. History of medical disease, which, in the opinion of the investigator, may put the participant at extra risk from study-related procedures or because disease may influence the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the UCSF Sinus Center practice of Drs. Andrew Goldberg and Steven Pletcher.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-01; Primary Completion 2017-09 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Severity of chronic rhinosinusitis as assessed by the Sino-Nasal Outcome Test-22 | 6 weeks following endoscopic sinus surgery
  This study enrolls participants with and without asthma with concomitant chronic rhinosinusitis (CRS). Investigators aim to study severity of CRS among the two groups following endoscopic sinus surgery. Severity of CRS will be judged using the Sino-Nasal Outcome Test-22, a paper-based, validated questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: John Fahy, MD, MSc, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Airway Clinical Research Center, San Francisco, California, United States